CLINICAL TRIAL: NCT00635362
Title: Immediate Post-placental Insertion of the Levonorgestrel-releasing Intrauterine System (LNG-IUS) After Cesarean Delivery vs. 4-8 Week Post-delivery Interval Insertion: A Randomized Controlled Trial
Brief Title: Postplacental Insertion of Levonorgestrel-releasing Intrauterine System (LNG-IUS) After Cesarean vs. Interval Insertion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15148A
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Contraception; Contraceptive Devices; Intrauterine Devices; Unplanned Pregnancy; Postpartum Period

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- postplacental insertion after cesarean (Experimental): Immediate postplacental insertion of the LNG-IUS through the uterine incision during cesarean, within 10 minutes after delivery of the placenta
  Device of intervention: Levonorgestrel-releasing intrauterine system (LNG-IUS)
  Interventions: Device: Levonorgestrel-releasing intrauterine system (LNG-IUS)
- delayed insertion group (Active Comparator): Insertion of the LNG-IUS 4-8 weeks after cesarean delivery
  Device of intervention: Levonorgestrel-releasing intrauterine system (LNG-IUS)
  Interventions: Device: Levonorgestrel-releasing intrauterine system (LNG-IUS)

INTERVENTIONS:
Device: Levonorgestrel-releasing intrauterine system (LNG-IUS) — Immediate postplacental insertion of the LNG-IUS through the uterine incision during cesarean, within 10 minutes after delivery of the placenta
  Other Names: Mirena IUD
  Arms: postplacental insertion after cesarean
Device: Levonorgestrel-releasing intrauterine system (LNG-IUS) — Insertion of the LNG-IUS 4-8 weeks after cesarean delivery
  Other Names: Mirena IUD
  Arms: delayed insertion group

SUMMARY:
The study is a randomized controlled trial comparing outcomes of immediate postplacental insertion of the levonorgestrel-releasing intrauterine system (LNG-IUS) vs. interval insertion of the LNG-IUS performed 4-8 weeks after delivery for patients undergoing scheduled cesarean delivery.

Our primary hypothesis is that the proportion of women using the LNG-IUS for contraception at 12 months after delivery will be higher in the group randomized to immediate post-placental insertion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at time of enrollment
* Planning to undergo a scheduled cesarean delivery
* Desires to use the LNG-IUS for contraception
* Willing and able to sign an informed consent in English
* Willing to comply with the study protocol
* Age greater than or equal to 18 years
* English speaking

Exclusion Criteria:

* Allergy to either polyethylene or levonorgestrel, or other contraindications to use of the LNG-IUS
* Positive testing for Gonorrhea, Chlamydia, or trichomoniasis during the pregnancy without treatment and a subsequent test of cure confirming a negative result
* Presence of leiomyomata significantly distorting the uterine cavity and thus not allowing placement of the LNG-IUS
* Uterine anomaly which would not allow placement of the LNG-IUS
* Current cervical cancer or carcinoma in-situ
* Desire for repeat pregnancy in less than 12 months
* History of postabortal or postpartum sepsis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Whitaker AK, Endres LK, Mistretta SQ, Gilliam ML. Postplacental insertion of the levonorgestrel intrauterine device after cesarean delivery vs. delayed insertion: a randomized controlled trial. Contraception. 2014 Jun;89(6):534-9. doi: 10.1016/j.contraception.2013.12.007. Epub 2013 Dec 26. PMID 24457061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Two urban academic medical centers from both pre-natal and Labor & Delivery clinics Dates: May 2007-January 2011 Inclusion: Pregnant, English-speaking women, aged 18 years and older, with planned cesarean delivery, and desiring the LNG-IUS were eligible for the study.
Groups:
- Delayed Insertion Group: Insertion of the LNG-IUS 4-8 weeks after cesarean delivery
  Device of intervention: Levonorgestrel-releasing intrauterine system (LNG-IUS)
  Levonorgestrel-releasing intrauterine system (LNG-IUS) : Insertion of the LNG-IUS 4-8 weeks after cesarean delivery
- Postplacental Insertion After Cesarean: Immediate postplacental insertion of the LNG-IUS through the uterine incision during cesarean, within 10 minutes after delivery of the placenta
  Device of intervention: Levonorgestrel-releasing intrauterine system (LNG-IUS)
  Levonorgestrel-releasing intrauterine system (LNG-IUS) : Immediate postplacental insertion of the LNG-IUS through the uterine incision during cesarean, within 10 minutes after delivery of the placenta
Period: Overall Study
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Started | 22 | 20
Completed | 9 | 12
Not Completed | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (5.3) | 27.1 (6.2) | 27.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42
Marital Status [Number; unit: participants]
  Single | 12 | 10 | 22
  Single, living with partner | 1 | 2 | 3
  Married | 9 | 8 | 17
Annual Income [Number; unit: participants]
  <$10,000 | 7 | 6 | 13
  $10,000-$30,000 | 6 | 7 | 13
  >$30,000 | 9 | 7 | 16
Insurance Coverage [Number; unit: participants]
  Medicaid | 16 | 14 | 30
  Private | 5 | 6 | 11
  Unknown/Not given | 1 | 0 | 1
Gestational Age at Delivery [Mean (Standard Deviation); unit: weeks] | 38.3 (1.7) | 38.4 (1.5) | 38.4 (1.6)
Parity at Enrollment [Number; unit: participants]
  0 | 1 | 1 | 2
  1 | 10 | 7 | 17
  2 | 8 | 9 | 17
  3 or more | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Use of the LNG-IUS for Contraception
Time Frame: 12 months after cesarean delivery
Measure: Number; unit: participants
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Number analyzed (Participants) | 22 | 20
participants
  Confirmed use of LNG-IUD | 9 | 12
  Lost to follow up at 12 months | 8 | 6
  Did not have IUD placed | 4 | 0
  Expelled prior to 12 months, not replaced | 0 | 2
  Removed per patient request | 1 | 0
Statistical Analysis 1: Comparison: Delayed Insertion Group vs Postplacental Insertion After Cesarean; Test type: Superiority or Other; p = 0.35, Fisher Exact

2. Secondary Outcome: Rates of Expulsion of the LNG-IUS
Time Frame: 12 months after cesarean delivery
Measure: Number; unit: participants
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Number analyzed (Participants) | 22 | 20
participants | 0 | 4
Statistical Analysis 1: Comparison: Delayed Insertion Group vs Postplacental Insertion After Cesarean; Test type: Superiority or Other; p = 0.04, Fisher Exact

3. Secondary Outcome: Perforation Rates
Time Frame: 12 months after cesarean delivery
Measure: Number; unit: participants
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Number analyzed (Participants) | 22 | 20
participants | 0 | 0
Statistical Analysis 1: Comparison: Delayed Insertion Group vs Postplacental Insertion After Cesarean; Test type: Superiority or Other; p = 1.000, Fisher Exact

4. Secondary Outcome: Satisfaction With LNG-IUS
Description: We measured satisfaction with the IUS at each visit using a single question with a 5 point Likert scale, with 1 being "very unsatisfied," 2 "unsatisfied", 3 "neutral," 4 "satisfied," and 5 "very satisfied." For statistical purposes, subjects were determined to be "SATISFIED" with the IUS if they chose either 4 or 5 for this question.
Time Frame: 6 months after cesarean delivery
Population: Analysis only done on subject completing six-month visit
Measure: Number; unit: participants
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Number analyzed (Participants) | 11 | 12
participants | 7 | 10
Statistical Analysis 1: Comparison: Delayed Insertion Group vs Postplacental Insertion After Cesarean; Test type: Superiority or Other; p = 0.37, Fisher Exact

5. Secondary Outcome: Satisfaction With LNG-IUS
Description: as for outcome 4
Time Frame: 12 months after cesarean delivery
Population: Analysis only done on subjects completing 12-month visit
Measure: Number; unit: participants
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Number analyzed (Participants) | 9 | 12
participants | 9 | 11
Statistical Analysis 1: Comparison: Delayed Insertion Group vs Postplacental Insertion After Cesarean; Test type: Superiority or Other; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Delayed Insertion Group | Postplacental Insertion After Cesarean
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 2/22 | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed Insertion Group (N=22) | Postplacental Insertion After Cesarean (N=20)
Chlamydia (Infections and infestations) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes